CLINICAL TRIAL: NCT02358122
Title: Determining the Potential of Wholegrain Wheat and Rye to Improve Gut HealTh
Acronym: RIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Lantmännens Forskningsstiftelse (Unknown)
Responsible Party: Principal Investigator, Mette Bredal Kristensen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-1-2014-062
Record Dates: First submitted 2015-01-21; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Gastrointestinal Diseases; Cardiovascular Diseases; Obesity
MeSH Terms: conditions — Gastrointestinal Diseases; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Refined wheat (Active Comparator): Refined wheat grain, a variety of cereal foods providing no wholegrain
  Interventions: Other: Refined wheat
- Wholegrain wheat (Experimental): Wholegrain wheat grain, a variety of cereal foods providing >100g wheat wholegrain/day
  Interventions: Other: Wholegrain wheat
- Wholegrain rye (Experimental): Wholegrain rye grain, a variety of cereal foods providing >100g rye wholegrain/day
  Interventions: Other: Wholegrain rye

INTERVENTIONS:
Other: Wholegrain rye — A variety of cereal foods providing >100g/day wholegrain from rye
  Arms: Wholegrain rye
Other: Wholegrain wheat — A variety of cereal foods providing >100g/day wholegrain from wheat
  Arms: Wholegrain wheat
Other: Refined wheat — A variety of cereal foods providing 0g/day wholegrain
  Arms: Refined wheat

SUMMARY:
A dietary intervention study designed as a randomized, controlled, parallel intervention of 6-weeks duration. A total of 75 participants will be included in the study and randomly allocated to one of three interventions (refined wheat, whoelgrain wheat or wholegrain rye). Clinincal examinations including anthropometric assessment, fecal, urine and fastign blood sampling, dietary assessment and a meal challenge will be done before (week 0) and after (week 6) the intervention. At timepoints week 0, 2, 4 and 6 questionnaires will be filled in concerning satisfaction with diet and gastrointestinal symptoms.

DETAILED DESCRIPTION:
A dietary intervention study designed as a randomized, controlled, parallel intervention of 6-weeks duration. A total of 75 participants will be included in the study and randomly allocated to one of three interventions (refined wheat, whoelgrain wheat or wholegrain rye). The randomization will be stratified according to sex and sex-specific median habitual cereal dietary fibre intake (16g/d for men and 13g/d for women). The randomization will be done by means of a randomization generator of the webpage (http://www.randomization.com). Recruitment and randomization will take place continuously during the study period, and therefore randomization will be done as mixed block randomization.

During the intervention study, participants are instructed to substitute all cereal products (e.g. bread, breakfast cereals, pasta) of their diet with the provided study products. The amount of provided study products will match the average intake of carbohydrate-rich products of the Danish population, which corresponds to ~200g of bread and cereal products per day. The participants will eat the study products in an ad libitum manner and b instructed to avoid other cereals in their diet including cake, biscuits, ready made meals and fast foods with the exception of White rice whis is allowed 1-2 times per week.

Clinincal examinations including anthropometric assessment, fecal, urine and fastign blood sampling, dietary assessment and a meal challenge will be done before (week 0) and after (week 6) the intervention. At timepoints week 0, 2, 4 and 6 questionnaires will be filled in concerning satisfaction with diet and gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 30 - 65 years

  * Body mass index (BMI): 25 - 32 kg/m2
  * Weight stable (<3 kg weight change during the last 6 months)
  * Apparently healthy
  * Informed consent signed
  * Freezer capacity for 2 weeks bread provision
  * Can attend all visits required for the study

Exclusion Criteria:

* • Smoking on a daily basis

  * Lactating (or lactating within 6 weeks prior to study start), pregnant (or pregnant within 3 months prior to study start) or wish to become pregnant during the study
  * Diagnosed with any form of diabetes or CVD
  * Reported chronic GI disorders
  * Antibiotic treatment 3 month before study start and during the study
  * Use of pre- or probiotic 1 month before study start and during the study
  * Lack of cooperation and adherence to the protocol
  * Use of prescription medication will be evaluated on an individual basis

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptoms evaluated by questionnaires (100mm visual analogue scales) | Change from 0 to 6 weeks
  Subjective sensations of gastrointestinal symptoms evaluated by questionnaires (100mm visual analogue scales)
Gut microbiota composition assessed using 16S in a single fecal sample | Change from 0 to 6 weeks
  Gut microbiota compostion assessed using 16S in a single fecal sample

SECONDARY OUTCOMES:
Anthropometric masures | Change from 0 to 6 weeks
  Body weight and waist circumference, saggital abdominal diameter and body composition (fat mass and fat free mass assessed using DEXA)
Blood pressure | Change from 0 to 6 weeks
  Diastolic and systolic blood pressure and heart rate assessed twice using an automated apparatus
Blood lipids, fasting concentrations of total, LDL and HDL cholesterol and triglyerides | Change from 0 to 6 weeks
  Fasting concentrations of total, LDL and HDL cholesterol and triglyerides
Glucose metabolism, fasting concentrations of glucose, insulin and HbA1C as calculation of HOMA-IR | Change from 0 to 6 weeks
  Fasting concentrations of glucose, insulin and HbA1C as calculation of HOMA-IR
Low-grade inflammation, fasting concentrations of hsCRP, IL-6, IL-10, and TNF-a | Change from 0 to 6 weeks
  Fasting concentrations of hsCRP, IL-6, IL-10, and TNF-a
Appetite sensation | Change from 0 to 6 weeks
  Fasting and postprandial (every 30 minutes for 240 minutes) sensation of hunger, satiety, fullness, prospective food intake, thirst and well being
Breath hydrogen assessed using a Hydrolyzer | Change from 0 to 6 weeks
  Fasting and postprandial (every 30 minutes for 240 minutes) concentrations of H2 in exhaled breath assessed using a Hydrolyzer
Short chain fatty acids, fecal concentrations of short chain fatty acids | Change from 0 to 6 weeks
  Fecal concentrations of short chain fatty acids
Fecal pH | Change from 0 to 6 weeks
  Fecal pH assessed in homogenized fecal sample
Intestinal permeability, assessed by urinary excretion of lactulose and mannitol | Change from 0 to 6 weeks
  Intestinal permeability is assessed by urinary excretion of lactulose and mannitol for 4 hours and 24 hours following an oral load of 10g lactulose and 2 g mannitol
Zonulin, fasting concentrations in plasma | Change from 0 to 6 weeks
  Fasting concentrations of zonulin in plasma
Dietary intake, a weighted 4-day food record | Change from 0 to 6 weeks
  a weighted 4-day food record will be used to assess energy intake and macronutrient (protein, fat, carbohydrates and dietaru fiber) composition
Compliance, measured by fasting plasma alkylresorcinol concentrations will be used as a biomarker of wholegrain wheat and rye intake | Change from 0 to 6 weeks
  Fasting plasma alkylresorcinol concentrations will be used as a biomarker of wholegrain wheat and rye intake

REFERENCES:
- [Derived] Christensen L, Vuholm S, Roager HM, Nielsen DS, Krych L, Kristensen M, Astrup A, Hjorth MF. Prevotella Abundance Predicts Weight Loss Success in Healthy, Overweight Adults Consuming a Whole-Grain Diet Ad Libitum: A Post Hoc Analysis of a 6-Wk Randomized Controlled Trial. J Nutr. 2019 Dec 1;149(12):2174-2181. doi: 10.1093/jn/nxz198. PMID 31504699
- [Derived] Vuholm S, Nielsen DS, Iversen KN, Suhr J, Westermann P, Krych L, Andersen JR, Kristensen M. Whole-Grain Rye and Wheat Affect Some Markers of Gut Health without Altering the Fecal Microbiota in Healthy Overweight Adults: A 6-Week Randomized Trial. J Nutr. 2017 Nov;147(11):2067-2075. doi: 10.3945/jn.117.250647. Epub 2017 Sep 27. PMID 28954842
- [Derived] Suhr J, Vuholm S, Iversen KN, Landberg R, Kristensen M. Wholegrain rye, but not wholegrain wheat, lowers body weight and fat mass compared with refined wheat: a 6-week randomized study. Eur J Clin Nutr. 2017 Aug;71(8):959-967. doi: 10.1038/ejcn.2017.12. Epub 2017 Mar 22. PMID 28327566